CLINICAL TRIAL: NCT05090033
Title: Secondary Use of Data Study Characterizing Kesimpta (Ofatumumab) Onboarding and Utilization in RMS Patients Using MSGo, With a Non-interventional Primary Use of Data Sub-study Comparing Patient Reported Outcomes Relative to Clinical Outcomes (EAFToS)
Brief Title: Characterizing the Use of Ofatumumab in a Real World Setting
Acronym: EAFToS
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GAU01
Record Dates: First submitted 2021-09-22; First posted 2021-10-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: ofatumumab; NIS; RMS
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Part I study cohort: Retrospective data analysis of up to 1500 de-identified participants contributing onboarding and adherence data via the MSGo Kesimpta Patient App.
  Interventions: Other: ofatumumab
- Part II study cohort: Up to 100 participants responding to PROs via the MSGo Patient App
  Interventions: Other: ofatumumab

INTERVENTIONS:
Other: ofatumumab — There is no treatment allocation. Patients administered ofatumumab by prescription that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This is a non-interventional primary use of data study utilizing de-identified patient-level onboarding and adherence data managed through the MSGo patient support service platform and includes a sub-study to explore the impact of ofatumumab on relevant patient reported outcomes (PROs) with respect to clinical outcomes.

DETAILED DESCRIPTION:
This study will be run in two parts. Part I will operate as a Secondary Use of Data study and Part II will operate as a Non-Interventional primary use of data study.

Part I: This study is descriptive in nature without any key underlying hypothesis and will explore the onboarding and adherence of RMS patients in Australia to ofatumumab treatment. De-identified patient-level onboarding and adherence data will be primarily generated and managed through the MSGo platform which will function as a Patient Support Service.

Part II: This part of the study will operate as a non-interventional primary use of data study and will explore the impact of ofatumumab on relevant patient reported outcomes (PROs) with respect to clinical outcomes. This part of the study will only be conducted at a selection of participating clinics. Patients in this part of the study will also have data collected as part of Part I of the study.

The data for the PROs will be collected through a mobile based application .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with relapsing forms of multiple sclerosis (RMS) to delay the progression of physical disability and reduce the frequency of relapse
* Expanded Disability Status Scale (EDSS) of 5.5 or lower (aligned with the plannedKEP criteria). Patients accessing ofatumumab through the PBS would have to meet the finalised restriction criteria (to be confirmed).
* Patients will provide consent to participate in Part I of the study through the MSGo experience program or patient support program onboarding process.
* Patients will need to provide additional consent to participate in Part II sub-study.

Exclusion Criteria:

* Patients diagnosed with Primary Progressive MS or Secondary Progressive MS without disease activity in line with the Australian Product Information].

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Australian patients with multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Part I and II: Proportion of doses not completed within three days of the expected date | Initiation
  Proportion of doses not completed within three days of the expected date during initiation to be collected
Part I and II: Proportion of doses not completed within 3 days of the expected date | First 3 months of maintenance
  Proportion of doses not completed within 3 days of the expected date during the first three months of maintenance to be collected

SECONDARY OUTCOMES:
Part I: Proportion of doses not completed within three days of the expected date | initiation period plus 12 months of maintenance
  Proportion of doses not completed within three days of the expected date to be collected
Part I: Proportion of doses not completed within 14 days of the expected date | 12 months of maintentance
  Proportion of doses not completed within 14 days of the expected date to be collected
Part I: Proportion of participants with a treatment interruption of more than six months during maintenance | Up to 18 months
  Proportion of participants with a treatment interruption of more than six months during maintenance to be collected.
  Interruption is calculated as 6 doses not completed
Part I: Proportion of participants discontinued within three months of the intial dose | Up to 18 months
  Proportion of participants discontinued within three months of the intial dose to be collected
Part I: Proportion of participants discontinued within 12 months of the intial dose. | Up to 18 months
  Proportion of participants discontinued within 12 months of the initial dose to be collected
Part I: Proportion of doses not completed within three days of the expected date for individual patient sub-groups | 12 months
  Patient sub-groups will be compared to either other complementary sub-groups or the "all patients" cohort
Part II: Proportion of doses not completed within 14 days of the expected date | during 18 months of maintenance
  This outcome measure will be measured for those patients who have MRI completed at approximately 18 months
Part II: proportion of participants discontinued within 18 months of the intial dose | within 18 months of the initial dose
  This outcome measure will be measured for those patients who have MRI completed at approximately 18 months
Part II: Change in work productivity measured by the Work Productivity and Activity Impairment (WPAI) questionnaire | Baseline,6 months, 12 months, 18 months
  The Work Productivity and Activity Impairment (WPAI) measures Four domain specific scores assessing work productivity and activity impairment (Absenteeism; Presenteeism; Mean work productivity; Activity impairment). Scores range from 0 to 100%. The four scores are expressed as impairment percentages with a higher score indicating less productivity and greater activity impairment.
Part II: Change in generic health status as measured by the EQ5D | Baseline, 6 months, 12 months, 18 months
  It comprises of a short descriptive system questionnaire and a visual analogue scale (VAS). The questionnaire provides a simple descriptive profile of a respondents health state and the VAS provides an alternative way to elicit an individuals rating of their own overall current health. Scale is rated from 0 (worst imaginable health) to 100 (the best imaginable scale)
Part II: Change in fatigue as measured by the Fatigue Scale for Motor and Cognitive Function (FSMC). | Baseline, 6 months, 12 months, 18 months
  The FSMC is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue).
Part II: Assessment of treatment satisfaction as measured by the Treatment Satisfaction Questionnaire for Medication (TSQM1.4) | Day 28, 6 months, 12 months, 18 months
  TSQM version 1.4 is a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. It comprises of 14 items assessing the following 4 domains: effectiveness (questions: 1-3), side effects (questions: 4-8), convenience (questions: 9-11), global satisfaction (questions: 12-14). For each of the 4 domains the scores of the corresponding items were added based on an algorithm to create a score of 0 to 100. Higher scores indicated greater satisfaction .
Part II: Proportion of self administration | 18 months
  Proportion of self administration as calculated by the number of self administered doses compared to the total number of doses over the total study time
Part II: Proportion of patients initiating ofatumumab who are treatment naïve | Baseline
  Proportion of patients initiating ofatumumab who are treatment naïve relative to prior high efficacy therapy as defined in Australia as alemtuzumab, ocrelizumab, natalizumab and cladribine) and other non-high efficacy Disease Modifying Therapies (DMTs).
Part II: Change in Expanded Disability Status Scale (EDSS) | Baseline, 6 months, 12 months
  EDSS is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS.
  EDSS scores range between 0 and 10 in 0.5 unit increments. Scores increase when the severity of the disability increases
Part II: Annualized relapse rate | 12 months
  Measured by number of relapses over a period of approximately 12 months.
Part II: Number of T1 Gd-enhancing lesions per MRI scan | Baseline, 6 months, 12 months
  This will only be assessed where gadolinium is used as per Institution's usual practice. Otherwise, this will not be reported
Part II: Number of new or enlarging T2 lesions on MRI | Baseline, 6 months, 12 months
  Number of new or enlarging T2 lesions on MRI to be collected
Percentage brain volume change | 12 months follow up
  The percent brain volume change analysis will be performed at 12 months follow up (either Month 12 (cf. Baseline) or Month 18 (cf. Month 6), via use of the SIENA method for atrophy analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Australia (7):
  - Novartis Investigative Site, Concord, New South Wales
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, St Leonards

IPD SHARING:
Plan to Share IPD: No